CLINICAL TRIAL: NCT03649828
Title: USE OF KEFIR AS A CO-ADJUVANT IN THE TREATMENT OF METABOLIC SYNDROME COMPONENTS: a Double-blind, Randomized, Placebo Controlled Clinical Trial
Brief Title: Kefir and Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Vila Velha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 43028115.8.0000.5064
Record Dates: First submitted 2018-05-02; First posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Metabolic Syndrome; Cardiovascular Diseases; Hypertension
Keywords: kefir; Probiotics; Metabolic Syndrome; Cardiovascular Diseases; Hypertension
MeSH Terms: conditions — Metabolic Syndrome; Cardiovascular Diseases; Hypertension | interventions — Kefir

STUDY DESIGN:
Intervention Model Description: There were two experimental groups. The kefir group (KG), that received orally probiotic milk fermented with the kefir grains, and the control group (CG), that received curd
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both Kefir and curd had been prepared to have the same consistency, color and flavor. Therefore, participants did not know if they were actually receiving kefir or curd. The care provider was a nutritionist that did not from each group the participants came from. There was two major investigators. The investigator responsible for the analysis of the data was also blind to the experimental groups, and he was also the outcome assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kefir group (Experimental): The kefir group (KG) received orally probiotic milk fermented with kefir grains and was compared with the control group (CG) that received only curd
  Interventions: Dietary Supplement: probiotic milk fermented with kefir grains
- control group (Experimental): control group (CG) that received only curd
  Interventions: Dietary Supplement: curd

INTERVENTIONS:
Dietary Supplement: probiotic milk fermented with kefir grains — Participants received probiotic milk fermented with kefir grains for consumption for 11 weeks. Before and after treatment, blood samples were collected for biochemical analysis and anthropometric data were also evaluated.
  Arms: kefir group
Dietary Supplement: curd — Participants received the curd for consumption for 11 weeks. Before and after treatment, blood samples were collected for biochemical analysis and anthropometric data were also evaluated.
  Arms: control group

SUMMARY:
Metabolic Syndrome (MS) contributes to the development of cardiovascular diseases (CVD). According to the World Health Organization (WHO), CVDs are the leading causes of death in the world. According to epidemiological data from the Ministry of Health, these diseases account for 29.4% of all deaths recorded in Brazil annually. Kefir is obtained by fermenting milk with kefir grains and has been recommended as a therapeutic form for the treatment of various clinical conditions. The hypothesis of the present study is that the daily intake of fermented beverages with kefir grains may reduce the risk factors associated with MS, thus reducing the incidence of CVD. A clinical trial was conducted with 48 volunteers, who presented at least three criteria for the diagnosis of MS. The subjects were divided into two groups that received for eleven weeks fermented dairy drink with kefir (KG) grains or homemade curd (CG). Weight and height measurements were taken to calculate BMI. The body composition evaluation was performed by determining the percentage of body fat and waist circumference (WC). The measurements of systolic blood pressure (SBP) and diastolic blood pressure (DBP) were taken. Blood samples were analyzed for fasting glycemia, glycated hemoglobin (HA1c), total cholesterol (TC), HDL cholesterol, triglycerides (Tg), C-reactive protein (CRP), aspartate aminotransferase (AST), Alanine Aminotransferase (ALT), Creatinophosphokinase (CPK), γ-Glutamyl Transferase (γ-GT), Urea Nitrogen, Urea and Creatinine. The level of non-HDL cholesterol (n-HDL) was determined by calculation. The Framingham score was used to assess the risk of developing cardiovascular events over the next ten years. Eleven weeks into the experiment, all measurements of body evaluation, SBP and DBP and biochemical analysis of blood were reevaluated.

DETAILED DESCRIPTION:
This is a randomized, double-blind clinical trial with stealth allocation through an automated randomization system Random Allocation Software version 1.0, May 2004. The randomization codes were the responsibility of the professional supervisor of the Laboratory of Technique and Dietetics of the University Vila Velha - UVV / ES. The same professional was responsible for the identification of bottled beverages intended for volunteers. Double blind refers to the blinding of patients, researcher, data collectors and outcome assessors. The kefir group (KG) received orally probiotic milk fermented with kefir grains and the control group (CG) received curds. The follow-up of the clinical trial is classified as long-term as it lasted for eleven weeks. The subjects of the research were recruited in an university teaching institution. After recruitment, confirmation of the presence of MS parameters was performed through anthropometric analyzes, blood pressure measurement and biochemical parameters, following the NCEP-ATP-III criteria. The subjects were then randomized into two groups, the control (CG) and kefir (KG). After the 11-week period all analyzes performed before the randomization process were repeated. During the study the drugs for the reduction of serum cholesterol, arterial hypertension and any other medication of continuous use had their use maintained. The inclusion criteria were age above 18 years and having had alteration of the components of MS. Pregnant and lactating women were excluded from the study, those who used drugs for dyslipidemias that interfered with intestinal metabolism such as ezetimibe and anion exchange resin, hormones of any kind, medicines for weight loss and the use of antioxidant supplements such as vitamin C or ω-3. The present work was submitted and approved by the Ethics Committee in Research with Human Subjects of the University Vila Velha - UVV, under number 1,025,083. All the volunteers signed the free and informed consent form, agreeing to participate in the research. The sample was calculated to detect a 12% reduction in the levels of ultra-sensitive C-reactive protein (CRP), considering a standard deviation of 15% a 2-tailed of 0.5 and power of 80%. The products were distributed to the volunteers in the workplace during office hours, in the morning, Monday to Friday. The routine was followed daily, totaling eleven weeks of experiment. The anthropometric measurements were individually assessed at the UVV Nutrition Clinic before the beginning of the trial and were repeated at the end of the study. In order to measure body weight, the RAMUZA DP-300 digital platform scale was used with a maximum capacity of 200 kg and a precision of 100 g. The measurements were performed with light clothing and with barefoot volunteers. The stature was measured using the CHORDER HM 210D digital vertical anthropometry, maximum measurement of 210 cm and precision of 1mm, with barefoot individuals. For the calculation and classification of the body mass index (BMI), the cuts proposed by the WHO were adopted. The waist circumference (WC) was obtained by means of a millimeter and inelastic measuring tape. The cut-off points for risk assessment associated with metabolic complications of obesity were proposed according to WHO and SIMÃO et al. (2013). Body composition was analyzed by electrical bioimpedance (MaltronBody Fat Analyzer BF 906), as described by Lukaski et al. (1985). The percentage of lean mass and body fat was evaluated. During the experiment the food selection was at the discretion of the volunteer, following the composition and distribution of the meals they usually consume. The blood pressure measurement (SBP and DBP) was performed according to the protocol of the Sixth Brazilian Hypertension Guideline, using the average between two measurements performed using HEM-705CPINT automatic device, Omron, OmronHealth Care, INC., Illinois-USA. For biochemical analysis, fasting blood samples were collected by traditional venipuncture to evaluate the biochemical parameters of fasting glycemia, glycated hemoglobin (HA1c), total cholesterol (TC), high density lipoprotein (HDLc), triglycerides (Tg) (C-reactive protein), C-reactive protein (CRP), low-oxidized lipoprotein (LDLox), Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Creatinophosphokinase (CPK), γ-Glutamyl Transferase (γ-GT), Urea Nitrogen, Creatinine. The samples were sent to the Tommasi Clinical Analysis Laboratory - Vila Velha - ES, for further analysis. Low Density Lipoprotein (LDLc) and Non-HDLc Cholesterol were calculated from the biochemical analysis of the blood. To identify the relative and absolute risk of each volunteer from the research for the development of coronary disease in the next decade of life, it was applied the Framingham score for the risk of coronary heart disease. All data from anthropometry, food intake, biochemical analysis of blood, SBP and DBP, and Framinghan score were collected before and after the period of consumption of curd or kefir products. The data was compiled in spreadsheet elaborated in Microsoft Excel and were expressed as the average plus or minus standard deviation (S.D.). The database was analyzed using the statistical program SPSS 11.5 (Statiscal Package Social Science version 11.5). Simple relative frequencies were performed for qualitative variables within each group. For the quantitative data, descriptive statistics were performed and the differences were determined using the paired Student's T test (in the same group) and unpaired (between the groups) for a 95% confidence interval. The difference between means will be considered when p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years, and;
* The presence of at least three of the five components of the metabolic syndrome.

Exclusion Criteria:

* Pregnant and lactating women;
* Subjects under the use of drugs for dyslipidemias that interfere with intestinal metabolism such as ezetimibe and anion exchange resin;
* Subjects under use of any kind of hormones;
* Subjects under the use of drugs for weight loss;
* Subjects under the use of antioxidant supplements such as vitamin C or ω-3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Ultra-sensitive C reactive Protein | 11 weeks
  Ultra-sensitive C reactive protein (uCRP) is a marker of cardiovascular risk. It is measured in blood samples and expressed in mg/dL. Therefore, the primary outcome was to evaluate the reduction of the cardiovascular risk. This measurement is stratified as bellow:
  Low cardiovascular risk: uCRP bellow 1.0 mg/dL; Medium cardiovascular risk: uCRP between 1.0 and 3.0 mg/dL; High cardiovascular risk: uCRP higher then 3.0 mg/dL.

SECONDARY OUTCOMES:
Framinghan score (the Coronay Heart Disease risk in 10 years) | 11 weeks
  The CHD (ten years risk) score is based on a group of variables: a) age, b) total cholesterol or Low disunity lipoprotein cholesterol, c) High density lipoprotein cholesterol, e) blood pressure, f) the presence of diabetes, and g) the smoke behavior. For each variable, the subject receives punctuation. Then, these punctuations are summed, and according with this sum a percentage of risk to develop CHD in 10 years is given.
  How much high is the sum, higher is the CHD risk. For men it varies from the sum ≤ -1, with the related CHD risk of 2%; to sum ≥14, with the related CHD risk ≥ 53%. For women it varies from the sum ≤ -1, with the related CHD risk of 1%; to sum ≥17, with the related CHD risk ≥ 27%.
  The calculation of this score (CHD risk in 10 yr) can be performed online and is based on the site of Framingham Heart Study. Therefore, the details of the process can be assessed in https://www.framinghamheartstudy.org/fhs-risk-functions/coronary-heart-disease-10-year-risk/.
Glycosylated hemoglobin | 11 weeks
  measurement of glycosylated hemoglobin in blood samples
Oxidized LDL-cholesterol | 11 weeks
  It has been considered a marker of development of atherosclerosis
Lipid profile | 11 weeks
  measurement of total cholesterol and fractions in the blood samples
Blood glucose | 11 weeks
  measurement of glucose and fractions in the blood samples
Blood pressure | 11 weeks
  indirect measurement of systolic and diastolic arterial pressure

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simao AF, Precoma DB, Andrade JP, Correa FH, Saraiva JF, Oliveira GM, Murro AL, Campos A, Alessi A, Avezum A Jr, Achutti AC, Miguel AC, Sousa AC, Lotemberg AM, Lins AP, Falud AA, Brandao AA, Sanjuliani AF, Sbissa AS, Alencar FA, Herdy AH, Polanczyk CA, Lantieri CJ, Machado CA, Scherr C, Stoll C, Amodeo C, Araujo CG, Saraiva D, Moriguchi EH, Mesquita ET, Fonseca FA, Campos GP, Soares GP, Feitosa GS, Xavier HT, Castro I, Giuliano IC, Rivera IV, Guimaraes IC, Issa JS, Souza JR, Faria NJ, Cunha LB, Pellanda LC, Bortolotto LA, Bertolami MC, Miname MH, Gomes MA, Tambascia M, Malachias MV, Silva MA, Izar MC, Magalhaes ME, Bacellar MS, Milani M, Wajngarten M, Ghorayeb N, Coelho OR, Villela PB, Jardim PC, Santos Filho RD, Stein R, Cassani RS, D'Avila RI, Ferreira RM, Barbosa RB, Povoa RM, Kaiser SE, Ismael SC, Carvalho T, Giraldez VZ, Coutinho W, Souza WK; Sociedade Brasileira de Cardiologia. [I Brazilian Guidelines for cardiovascular prevention]. Arq Bras Cardiol. 2013 Dec;101(6 Suppl 2):1-63. doi: 10.5935/abc.2013S012. No abstract available. Portuguese. PMID 24554026
- [Background] National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) final report. Circulation. 2002 Dec 17;106(25):3143-421. No abstract available. PMID 12485966
- [Background] Kumar M, Nagpal R, Kumar R, Hemalatha R, Verma V, Kumar A, Chakraborty C, Singh B, Marotta F, Jain S, Yadav H. Cholesterol-lowering probiotics as potential biotherapeutics for metabolic diseases. Exp Diabetes Res. 2012;2012:902917. doi: 10.1155/2012/902917. Epub 2012 May 3. PMID 22611376
- [Background] Labonte ME, Dewailly E, Lucas M, Couture P, Lamarche B. Association of red blood cell n-3 polyunsaturated fatty acids with plasma inflammatory biomarkers among the Quebec Cree population. Eur J Clin Nutr. 2014 Sep;68(9):1042-7. doi: 10.1038/ejcn.2014.125. Epub 2014 Jul 16. PMID 25028086
- [Background] Friques AG, Arpini CM, Kalil IC, Gava AL, Leal MA, Porto ML, Nogueira BV, Dias AT, Andrade TU, Pereira TM, Meyrelles SS, Campagnaro BP, Vasquez EC. Chronic administration of the probiotic kefir improves the endothelial function in spontaneously hypertensive rats. J Transl Med. 2015 Dec 30;13:390. doi: 10.1186/s12967-015-0759-7. PMID 26715471
- [Background] Lukaski HC, Johnson PE, Bolonchuk WW, Lykken GI. Assessment of fat-free mass using bioelectrical impedance measurements of the human body. Am J Clin Nutr. 1985 Apr;41(4):810-7. doi: 10.1093/ajcn/41.4.810. PMID 3984933
- [Background] Pearson TA, Mensah GA, Alexander RW, Anderson JL, Cannon RO 3rd, Criqui M, Fadl YY, Fortmann SP, Hong Y, Myers GL, Rifai N, Smith SC Jr, Taubert K, Tracy RP, Vinicor F; Centers for Disease Control and Prevention; American Heart Association. Markers of inflammation and cardiovascular disease: application to clinical and public health practice: A statement for healthcare professionals from the Centers for Disease Control and Prevention and the American Heart Association. Circulation. 2003 Jan 28;107(3):499-511. doi: 10.1161/01.cir.0000052939.59093.45. No abstract available. PMID 12551878